CLINICAL TRIAL: NCT05433623
Title: Vascular Surgery Admissions in a Tertiary Care Hospital in the Mid-West: A 12 Month Profile.
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient resources to complete this project.
Sponsor: University Hospital of Limerick (Other)
Responsible Party: Principal Investigator, Fiona Leahy, Research Nurse Manager, University Hospital of Limerick
Other Study IDs: DVS001
Record Dates: First submitted 2022-06-01; First posted 2022-06-27 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Vascular Surgery Admissions: Patients who present and/or are admitted to University Hospital Limerick under the care of a Vascular Consultant.
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — It will be documented if the patient underwent surgery for their vascular issue

SUMMARY:
Creating a 12 month profile of Vascular Surgery Admissions aims to inform service delivery and optimise patient care resources. There is a gap in the literature pertaining to this topic, particularly from an Irish perspective. This research could inform a clinical pathway to reduce LOS for patients cared for by the Department of Vascular Surgery.

DETAILED DESCRIPTION:
This is an observational cross sectional study. This study will be mixed methods. Following the profile creation the researcher aims to complete qualitative research in the form of interviewing a cohort of vascular patients about their experiences in order to inform practice development. Ethics approval will be granted prior to any activities taking place.

Selection/Recruitment:

Patients attending UHL deemed to have vascular care needs and assigned to the care of a Vascular Consultant will be included in this study. The data will be collected 12 months from the date of commencing the study. Vascular consults will be excluded for the purpose for this research unless care is transferred. Informed consent is not required for this research so there in no exclusion criteria in relation to ability to provide same.

Data Collection:

The data to inform this project will be collected from medical chart review and utilising the UHL inpatient IT systems. No patient identifiers will be collected for this research and it will comply with GDPR. The Ipims system will be used to measure current inpatients under the care of a Vascular Consultant. HIPE data will be requested to examine the length of stay for vascular inpatients. The individual's medical notes will be reviewed to assess:

* Reason for admission to hospital and/or presentation to the Emergency Department (ED).
* Date, day and time of admission.
* Referral source.
* Categorisation from triage in the ED if applicable.
* Consultant caring for the individual.
* Demographic profile & Brief Medical and Surgical History.
* ? Elective or Emergency admission.
* ? Intervention or conservative management. Treatment course.
* ? Re-admission.
* Length of stay.
* Time patient waited for theatre procedure (date of admission to date of theatre) including fasting time.
* Time patient waited for vascular scans (date of admission to date of scans) & scans completed.
* Time patient waited for rehab (transfer) if applicable.
* Time patient waited for OPAT if applicable.
* Clinical Frailty Scale (Appendix II) & Charlson Co-Morbidity Scale (Appendix III) (no patient intervention required).

Data Analysis:

Descriptive statistics with multivariant analyses.

Process Evaluation:

The MRC Framework will be employed for process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending UHL deemed to have vascular care needs and assigned to the care of a Vascular Consultant will be included in this study.
* The data will be collected 12 months from the date of commencing the study.

Exclusion Criteria:

* Patients outside of the set dates will be excluded.
* Vascular consults will be excluded for the purpose of this research unless care is transferred.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study aims to create a profile f vascular admissions to a tertiary care hospital in the Mid West of Ireland and describe the characteristics of the admission.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Clinical Frailty Scale | 1 year
  Clinical frailty score will be determined for vascular patient admissions. This is a 9 point scale. the higher the score means the greater the risk.
Charlson Co-Morbidity Scale | 1 year
  Scoring will be determined for vascular patient admissions. The Charlson Comorbidity Index (CCI) assesses comorbidity level by taking into account both the number and severity of 19 pre-defined comorbid conditions. It provides a weighted score of a client's comorbidities which can be used to predict short term and long-term outcomes such as function, hospital length of stay and mortality rates.
Admission details | 1 year
  Length of stay, interventions, referral source will be documented

IPD SHARING:
Plan to Share IPD: No
The researcher will not be sharing IPD